CLINICAL TRIAL: NCT03402061
Title: Nutrition in Disguise: Improving the Nutritional Quality of Foods for Older Adults
Brief Title: Nutrition in Disguise: Development and Palatability Testing of Novel Food Products
Acronym: NiD
Status: Completed | Type: Observational
Sponsor: University of Waterloo (Other)
Collaborators: The Weston A. Price Foundation (Other); University of Guelph (Other)
Responsible Party: Principal Investigator, Heather Keller, Principal Investigator, University of Waterloo
Other Study IDs: ORE22605
Record Dates: First submitted 2018-01-01; First posted 2018-01-17 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Community living seniors: Approximately 50 seniors will taste test each nutrient enhanced recipe and determine acceptability and palatability.
  Interventions: Dietary Supplement: nutrient enhanced recipes
- LTC cognitively well: Approximately 15 seniors living in long term care who do not have cognitive impairment will taste test each nutrient enhanced recipe and determine acceptability and palatability.
  Interventions: Dietary Supplement: nutrient enhanced recipes
- LTC persons living with dementia: Approximately 15 seniors living in long term care with cognitive impairment will taste test each nutrient enhanced recipe and determine acceptability and palatability.
  Interventions: Dietary Supplement: nutrient enhanced recipes

INTERVENTIONS:
Dietary Supplement: nutrient enhanced recipes — normal ingredients will be substituted to promote nutrient density of products

SUMMARY:
Nutrition in Disguise is focused on developing and testing the acceptability of nutrient dense food products appropriate for older adults and specifically those living in long term care.

DETAILED DESCRIPTION:
Project Description: The overall goal of this research is to develop food recipes that are rich in vitamins, minerals and other food components known to support the physical and mental health of older adults. A variety of enhanced food recipes will be initially designed for older adults living in residences with applicability to pre-frail and frail older adults living in the community. It is hypothesized that the nutrient (protein and vitamins and minerals) density and anti-oxidant (i.e. phytochemical) potential of menus used in residential environments can be improved in a cost-effective manner with the inclusion of several enhanced food recipes designed for this population. This will be achieved by identifying high nutrient ingredients that can be incorporated into recipes of foods that are highly consumed by this segment. Initial work will summarize what is known from existing literature about micronutrient deficiencies and interventions with vitamins, minerals and antioxidants to improve the health of older adults. Foods commonly consumed that can be enhanced to promote their nutritional density (e.g. more nutrients in less calories) will be identified and recipes developed and tested with older adults living in the community and in residences. Products that pass this testing will then be introduced into a residence menu rotation to determine if they are well accepted by residents. A cost benefit of introducing these new products into a residence menu will be demonstrated by showing the gains in nutritional quality of the menu for the cost of producing these products in the home.

Relevance to the field of food innovation: Currently, older adults, especially those who are frail or live in residences, do not consume adequate nutrition to optimize their health. Micronutrient inadequacies are a potential problem. Research to date suggests that diet can also be supportive for delaying frailty and slowing the progression of dementia. Yet, food choices and offerings can be low in nutrition. Cost effective, innovative recipes that used common ingredients to reach nutrition goals for older adults are needed.

Anticipated outcomes:

Up to 10 enhanced recipes that have been developed for residences will be developed and tested for palatability. Knowledge tools will be created for home chefs on how to incorporate nutrient dense ingredients into recipes and how to use the information gained in this project for menu planning.

ELIGIBILITY:
Inclusion Criteria:

* Older adults living in the community with no food allergies
* older adults living in long term care with and without dementia with no food allergies

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Approximately 50 community living seniors will test each product. 15 senior residents with and 15 without dementia will be recruited as a 'taste test panel' from long germ care homes
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Palatability Scale | 19 months
  Participants rate the palatability of the enhanced recipe sample using a five point scale (liked very much to disliked very much) with questions on flavour, texture, appearance, overall liking and ask if the participant woudl eat this product again

CONTACTS AND LOCATIONS:
Overall Officials: Heather Keller, PhD, Principal Investigator — University of Waterloo
Locations (1):
- Research Institute for Aging, Waterloo, Canada

IPD SHARING:
Plan to Share IPD: No